CLINICAL TRIAL: NCT00798941
Title: ICU Patient and Family Comfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Palliative Care Research Center (Other)
Responsible Party: Kathleen Puntillo, U.C. San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08033609
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-06

CONDITIONS: Pain; Thirst; Anxiety; Satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction | interventions — Oral Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pain intervention (Experimental): music and massage for 30 minutes
  Interventions: Behavioral: pain intervention
- thirst intervention (Experimental): sterile water mouth spray, lip moisturizer,mouth swab
  Interventions: Behavioral: mouth care
- control (No Intervention)

INTERVENTIONS:
Behavioral: mouth care — mouth spray, mouth swab, moisturizer
  Arms: thirst intervention
Behavioral: pain intervention — music and massage
  Arms: pain intervention

SUMMARY:
The purpose of this study is to evaluate family-led interventions for Intensive Care Unit (ICU) patients' symptoms (i.e., pain and thirst) that will involve ICU patients' family members in the non-pharmacological management of these symptoms. This family involvement may help to ameliorate not only patients' symptoms but also the families' symptoms and promote family satisfaction with ICU care.

ELIGIBILITY:
Inclusion Criteria:

* Patient:

  * in ICU for at least 24 hours;
  * adult;
  * able to self-report;
  * pain and thirst greater than 3 on 0-10 numeric rating scale;
  * English-speaking.
* Family member:

  * 18 years or older;
  * visits patient more than other family members;
  * closest person to patient (can be non-biological).

Exclusion Criteria:

* Patient:

  * in ICU for at less than 24 hours;
  * non-adult;
  * unable to self-report;
  * no pain and thirst greater than 3 on 0-10 numeric rating scale;
  * non-English-speaking.
* Family member:

  * younger than 18 years;
  * visits patient less than other family members;
  * not closest person to patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
patient-reported pain | immediately after intervention

SECONDARY OUTCOMES:
patient-reported thirst | immediately after intervention
Family-reported anxiety | at end of study
Family-reported satisfaction | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Puntillo, DNSc, Principal Investigator — U.C. San Francisco
Locations (1):
- U.C. San Francisco, San Francisco, California, United States